CLINICAL TRIAL: NCT03069911
Title: Randomized Controlled Trial of OnabotulinumtoxinA for Depression in Parkinson Disease
Brief Title: Trial of OnabotulinumtoxinA for Depression in Parkinson Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit required participants
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00082708
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease; Depression
Keywords: Parkinson Disease; Parkinsonism; Depression; OnabotulinumtoxinA; BOTOX
MeSH Terms: conditions — Parkinson Disease; Depression; Parkinsonian Disorders | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): One injection of onabotulinumtoxinA (29 units for women and 40 units for men) will be injected into two facial muscles - the corrugator and procerus.
  Interventions: Biological: OnabotulinumtoxinA
- Control (Placebo Comparator): One injection of saline solution will be injected into two facial muscles - the corrugator and procerus.
  Interventions: Biological: Control

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA (29 units for women; 40 units for men) diluted with 0.9% sodium chloride (saline) solution to 40 units per milliliter (mL) (0.725 mL for women, 1 mL for men)
  Other Names: Botox; Botulinum Toxin Type A
  Arms: Intervention
Biological: Control — 0.9% sodium chloride solution (saline) solution injections (0.725mL for women, 1mL for men)
  Other Names: Normal saline
  Arms: Control

SUMMARY:
This study evaluates the efficacy of onabotulinumtoxinA (BOTOX®) in the treatment of depression associated with Idiopathic Parkinson Disease in adults. As a Randomized Controlled Trial, half of the participants will receive onabotulinumtoxinA injections and half will receive a placebo saline solution.

DETAILED DESCRIPTION:
Depression is a common, but treatable, comorbid condition often seen in persons with Idiopathic Parkinson Disease (iPD). Depression in Parkinson Disease may be hard to treat as patients with iPD may be sensitive to side effect of medication. As a result, other treatments which have better side effects profiles than antidepressants may be equivalent (or better) options.

OnabotulinumtoxinA is a purified formulation of botulinum toxin serotype A which is widely utilized for neurological (and cosmetic) purposes in medicine. OnabotulinumtoxinA has preliminary studies showing it may be beneficial for the treatment of Major Depressive Disorder when given in isolated injections to facial muscles (corrugator and procerus). When given in low doses, onabotulinumtoxinA is thought to have minimal side effects.

The investigators propose that a single treatment onabotulinumtoxinA may improve symptoms of depression in persons with Parkinson Disease over three months compared to placebo. The investigators plan to use both subjective and objective evaluations of depression symptoms and regular physical exams to ensure physical (motor) symptoms of Parkinson Disease do not worsen.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained in the English language;
* They are a 18 to 95 years old;
* They meet United Kingdom Brain Bank Criteria for probable idiopathic Parkinson disease;
* They meet Diagnostic and Statistical Manual (DSM)-IV criteria for major depressive disorder (MDD) as diagnosed by the M.I.N.I. at screening;
* They are judged by the investigator to have the capacity to understand the nature of the study;
* They are willing to comply with all the requirements of the study;
* They are considered by the investigator to be likely to adhere to the protocol.

Exclusion Criteria:

* They have been treated with onabotulinumtoxinA injected into the facial muscles for any reason in the 3 months prior to screening;
* They have Bipolar Disorder, Post-Traumatic Stress Disorder, a Psychotic Disorder or any other non-unipolar depressive disorder as a principal diagnosis in the 6 months prior to screening;
* They endorse active suicidal ideation at enrollment or during any study visit, or have attempted suicide in the six months prior to screening;
* They have a history of substance abuse or dependence in the 2 months prior to screening;
* They test positive for illicit drugs on urine screen, and this has not been adequately explained to the satisfaction of the investigator
* They are considered to be at significant risk of committing homicide;
* They have an unstable medical condition;
* Women of childbearing potential who are pregnant or are considering becoming pregnant during the length of the study;
* There has been a change in their PD medication or psychotherapy treatment regimen in the 30 days preceding screening;
* They are regarded, for any reason, by the principal investigator as being an unsuitable candidate for the protocol.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HDRS) | Baseline and two visits over three months (weeks 6 and 12)
  Improvement on a clinician-rated objective scale for depression as assessed over two weeks (6 weeks and 12 weeks after treatment)
Clinical Global Impression - Improvement (CGI-I) | Baseline and two visits over three months (weeks 6 and 12)
  Improvement on a measure of global change from screening to study discontinuation
Clinical Global Impression - Severity (CGI-S) | Baseline and two visits over three months (weeks 6 and 12)
  Improvement on measure of global illness severity from screening to study discontinuation
Beck Depression Inventory II | Baseline and two visits over three months (weeks 6 and 12)
  Improvement on a participant-rated subjective scale for depression as assessed over two visits

SECONDARY OUTCOMES:
Clinical Severity Score for Glabellar Frown Lines | Baseline and two visits over three months (weeks 6 and 12)
  Assessment of change in participant frowning before and after onabotulinumtoxinA injections and relationship with depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Pantelyat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified group data will be shared between the two study sites (Johns Hopkins and NIH)